CLINICAL TRIAL: NCT06502587
Title: Effects of Blood Flow Restriction Training With Low Intensity Exercises on Pain,Range of Motion and Quality of Life in Knee Osteoarthritis
Brief Title: Effects of Blood Flow Restriction Training With Low Intensity Exercises in Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/01112
Record Dates: First submitted 2024-06-11; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Knee Osteoarthritis
Keywords: Blood flow restriction training; Knee Osteoarthritis; Pain; Quality of life; Range of motion
MeSH Terms: conditions — Osteoarthritis, Knee; Pain | interventions — Blood Flow Restriction Therapy; Ultrasonic Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- blood flow restriction training (Experimental): we will apply blood flow restriction training with low intensity exercises on patients with knee osteoarthritis to check pain,quality of life and range of motion.
  Interventions: Other: blood flow restriction training
- ultrasound application only (Active Comparator): in this group we will apply ultrasound therapy on knee joint for 7 minutes.
  Interventions: Other: ultrasound therapy

INTERVENTIONS:
Other: blood flow restriction training — we will apply blood flow restriction training with low intensity exercises like knee flexion ,knee extension and straight leg raise 10 repetitions 2 sets a day and 3 times/week a rest interval of 2 minutes between exercises, for 30 minutes of this whole procedure.
  total 12 sessions given in 4 weeks each session of maximum 30 minutes
  Arms: blood flow restriction training
Other: ultrasound therapy — All subjects will be given Ultrasound therapy as per patient requirement with 1.5 Watts/cm^2 in continuous mode around knee joint. Conservative exercises(quads isometric exercise, pillow squeeze, heel raise, straight leg raise and side leg raise) will be applied for 3 times per week (daily one set of 10 repetitions) They will be given this treatment for 3 times per week
  Arms: ultrasound application only

SUMMARY:
The aim of the study is to examine the effects of blood flow restriction training(BFRT) with low intensity exercises on pain, range of motion and quality of life in Knee Osteoarthritis. A randomized clinical trial will be conducted at Lahore general hospital. Non-probability convenience sampling will be used, and 36 subjects, age 40-65 years will be randomly allocated into two groups by lottery method after meeting the inclusion criteria.

DETAILED DESCRIPTION:
The aim of the study is to examine the effects of blood flow restriction training(BFRT) with low intensity exercises on pain, range of motion and quality of life in Knee Osteoarthritis. A randomized clinical trial will be conducted at Lahore general hospital. Non-probability convenience sampling will be used, and 36 subjects, age 40-65 years will be randomly allocated into two groups by lottery method after meeting the inclusion criteria. Both groups will receive Ultrasound therapy for 7 minutes, as common treatment. Group A will be treated with Blood flow restriction training with low intensity exercises and Group B will be treated with baseline treatment only. 3 sessions per week and total 12 sessions for 4 weeks. The outcome measures will be conducted through NPRS, Womac index for osteoarthritis,kellgren and lawrence scale and goniometry before and after 4 weeks. Data will be analyzed using SPSS software version 26.

ELIGIBILITY:
Inclusion Criteria:

* Both Male and Female age between 40 to 65 years diagnosed with womac ostearthritis index having acute knee pain.
* Patients with history of osteoarthritis (of grade 1 and 2 with KL(kellgren and Lawerence)) grading system for knee Osteoarthritis
* Pain in and around knee measuring through Numeric Pain rating Scale(NPRS)>4(14)

Exclusion Criteria:Patient with history of

* hypertension
* diabetes
* sickle cell anemia
* renal compromise
* obesity
* open fracture,
* increased intracranial pressure
* pregnancy
* cancer or tumor,
* extremity with dialysis access,
* extremity fracture
* peripheral vascular compromise
* DVT(Deep vein thrombosis) & pulmonary embolism deformity of hip & back

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-11-23 (Actual); Primary Completion 2024-07-20 (Estimated); Study Completion 2024-07-20 (Estimated)

PRIMARY OUTCOMES:
NPRS Numeric pain rating scale | 4th week
  The NPRS is a self-reported, or clinician administered, measurement tool consisting of a numerical point scale with extreme anchors of 'no pain' to 'extreme pain'. The scale is typically set up on a horizontal or vertical line, ranges most commonly from 0-10 or 0-100, and can be administered in written or verbal form. The patient is asked to rate his/her pain intensity and a particular time frame or descriptor is established (e.g. within the last 24 h, today, worst pain, average pain, or least pain)

SECONDARY OUTCOMES:
Womac index for knee osteoarthritis | 4th week
  WOMAC measures three separate dimensions: Pain (5 questions), Stiffness (2 questions), and Pain, stiffness, and physical function were measured by WOMAC. This instrument is validated and recommended by the Osteoarthritis Research Society as the measure of choice when assessing health status in older adults with knee OA. Rating scale ranges from 0 (none) to 4 (extreme), with higher total scores indicating greater dysfunction.The WOMAC addresses symptoms and functional disability in separate scales . Also, the WOMAC is a patient questionnaire.
Knee Related QOL (QUALITY OF LIFE) Subscale From KOOS | 4th week
  The Knee injury and Osteoarthritis Outcome Score (KOOS) was developed as an extension of the WOMAC Osteoarthritis Index with the purpose of evaluating short-term and long-term symptoms and function in subjects with knee injury and osteoarthritis The KOOS holds five separately scored subscales: Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related Quality of Life (QOL). The effect size is generally largest for the subscale QOL followed by the subscale Pain. The KOOS is a valid, reliable and responsive self-administered instrument that can be used for short-term and long-term follow-up of several types of knee injury including osteoarthritis
Universal goniometer | 4th week
  The most common tool for measuring ROM has been the universal goniometer (UG; full-circle manual goniometer. The advantage with the UG is its low cost, but both hands are needed to perform the measurements

CONTACTS AND LOCATIONS:
Overall Officials: Iqra Khan, Mphil, Principal Investigator — Riphah International University
Locations (1):
- Lahore General Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prathap Kumar J, Arun Kumar M, Venkatesh D. Healthy gait: Review of anatomy and physiology of knee joint. International Journal of Current Research and Review. 2020;12(6):1-8.
- [Background] Van Cant J, Dawe-Coz A, Aoun E, Esculier JF. Quadriceps strengthening with blood flow restriction for the rehabilitation of patients with knee conditions: A systematic review with meta-analysis. J Back Musculoskelet Rehabil. 2020;33(4):529-544. doi: 10.3233/BMR-191684. PMID 32310159
- [Background] Ferlito JV, Pecce SAP, Oselame L, De Marchi T. The blood flow restriction training effect in knee osteoarthritis people: a systematic review and meta-analysis. Clin Rehabil. 2020 Nov;34(11):1378-1390. doi: 10.1177/0269215520943650. Epub 2020 Aug 10. PMID 32772865
- [Background] Ferraz RB, Gualano B, Rodrigues R, Kurimori CO, Fuller R, Lima FR, DE Sa-Pinto AL, Roschel H. Benefits of Resistance Training with Blood Flow Restriction in Knee Osteoarthritis. Med Sci Sports Exerc. 2018 May;50(5):897-905. doi: 10.1249/MSS.0000000000001530. PMID 29266093
- [Background] Grantham B, Korakakis V, O'Sullivan K. Does blood flow restriction training enhance clinical outcomes in knee osteoarthritis: A systematic review and meta-analysis. Phys Ther Sport. 2021 May;49:37-49. doi: 10.1016/j.ptsp.2021.01.014. Epub 2021 Feb 3. PMID 33582442
- [Background] Kaya PDCBK, Alpozgen AZ. EFFECTS OF BLOOD FLOW RESTRICTION METHOD IN KNEE PATHOLOGIES. TAM METİN KİTABI. 2022:21.
- [Background] Wang HN, Chen Y, Cheng L, Cai YH, Li W, Ni GX. Efficacy and Safety of Blood Flow Restriction Training in Patients With Knee Osteoarthritis: A Systematic Review and Meta-Analysis. Arthritis Care Res (Hoboken). 2022 Jan;74(1):89-98. doi: 10.1002/acr.24787. Epub 2021 Dec 17. PMID 34549541
- [Background] Pitsillides A, Stasinopoulos D, Mamais I. Blood flow restriction training in patients with knee osteoarthritis: Systematic review of randomized controlled trials. J Bodyw Mov Ther. 2021 Jul;27:477-486. doi: 10.1016/j.jbmt.2021.04.015. Epub 2021 Apr 23. PMID 34391274
- [Background] Li S, Shaharudin S, Abdul Kadir MR. Effects of Blood Flow Restriction Training on Muscle Strength and Pain in Patients With Knee Injuries: A Meta-Analysis. Am J Phys Med Rehabil. 2021 Apr 1;100(4):337-344. doi: 10.1097/PHM.0000000000001567. PMID 33727516
- [Background] Mahmoud WS, Osailan A, Ahmed AS, Elnaggar RK, Radwan NL. Optimal parameters of blood flow restriction and resistance training on quadriceps strength and cross-sectional area and pain in knee osteoarthritis. Isokinetics and Exercise Science. 2021;29(4):393-402.
- [Background] NADIA AF, ABDALLAH MM, FADEL MEM, MOHAMMED MM. Effect of Low Load Resistance Blood Flow Restriction Training on Knee Osteoarthritis. The Medical Journal of Cairo University. 2018;86(December):4297-306.
- [Background] Rolff S, Korallus C, Hanke AA. [Rehabilitation with the aid of blood flow restriction training]. Unfallchirurg. 2020 Mar;123(3):180-186. doi: 10.1007/s00113-020-00770-1. German. PMID 32030478